CLINICAL TRIAL: NCT06912568
Title: Three-dimensional CBCT Analysis of Root Volume Changes Following Tooth-bone and Bone-borne Maxillary Expansion: A Pilot Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Michele Cassetta, Full Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URomLS_5951a
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Root Resorption; Orthodontic Appliance; CBCT Segmentation
Keywords: tooth-borne RME; bone-borne RME; external root resorption; maxillary expansion; CBCT; miniscrews
MeSH Terms: conditions — Root Resorption | interventions — Tissue Expansion Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 4 miniscrews Bone-borne expansion group (Experimental)
  Interventions: Device: Miniscrew insertion; Device: Expander; Radiation: CBCT
- 2 miniscrews bone-borne group (Experimental)
  Interventions: Device: Miniscrew insertion; Device: Expander; Radiation: CBCT
- tooth-borne expander (Experimental)
  Interventions: Device: Expander; Radiation: CBCT

INTERVENTIONS:
Device: Miniscrew insertion — four or two miniscrews insertions using computer-guided minimally-invasive and flapless approach
  Arms: 2 miniscrews bone-borne group; 4 miniscrews Bone-borne expansion group
Device: Expander — In the TB group, the tooth-borne hyrax appliance was designed with bands on the maxillary first molars; in the BB4 group, the bone-borne expander was supported by 4 miniscrews inserted both in paramedian and parapalatal position of the palatal vault; in the BB2 group, the bone-borne expander was supported by 2 miniscrews inserted in the paramedian region of the palate. The same type of expansion screw and expansion protocol were used in all groups. Specifically, a 10mm hyrax click screw (Dentaurum, Bologna, Italy) was activated by 4 quarter-turns on the first day and by 3 quarter-turns per day during the active phase of treatment (0.20mm per turn, 0.6mm daily) until an 8mm screw opening was achieved.
Radiation: CBCT — All patients underwent CBCT examinations before the application of the RME device (T0) and post-treatment, after the 6-month retention period (T1). The exposure settings were as follows: 10 mA, 90 kV, total scanning time of 15.0 seconds, effective radiation time of 4.0 seconds, voxel size of 0.2 mm, scanning area of 14 x 16.5 cm, and an effective radiation dose of approximately 524 mGy/cm2.
  The CBCT images analyzed in this study were not acquired specifically for this research but were part of an ongoing prospective randomized clinical trial aimed at evaluating the skeletal and dentoalveolar effects of three different orthodontic devices. The imaging protocol was established in accordance with ethical guidelines and was approved by the relevant institutional review board.

SUMMARY:
External root resorption (ERR) is an undesired side effect observed after rapid maxillary expansion (RME). This study aimed to investigate changes in the root volume of maxillary permanent first molars after RME using tooth-borne and bone-borne devices with cone-beam computed tomography (CBCT) software analysis.

The study included 21 patients (mean age 11.8 years ±0.79 years) with skeletal transverse maxillary deficiency, randomly allocated into three groups according to the type of expansion device: tooth-borne Hyrax (TB), bone-borne 4-miniscrew (BB4) and bone-borne 2-miniscrew (BB2). The same expansion screw and activation protocol were applied in all groups. A CBCT was carried out before treatment (T0) and after treatment at a 6-month follow-up (T1). The volumetric assessment of maxillary permanent first molars was performed using digital software, evaluating the mean root volume changes (mm3 and %) between T0 and T1 in each group (TB, BB4, BB2). The Wilcoxon test was used for intra-group comparisons and the Kruskal-Wallis test was used for inter-group comparisons. Significance was set at P≤0.05.

DETAILED DESCRIPTION:
Significant forces are transmitted to the maxilla through the anchored teeth in tooth-borne maxillary expansion. Despite the clinical therapeutic benefits that may be achieved, this treatment is not without drawbacks. Tooth-anchored appliances have been associated with several adverse effects on the teeth and surrounding tissues, including reduced buccal bone thickness, bone fenestration, gingival recession, and root resorption (RR). Root resorption can be defined as a physiologic or pathologic condition resulting in the dissolution of the cementum and dentin of dental roots and may represent an inevitable consequence of orthodontic treatment and active tooth movement. In this regard, a systematic review by Lo Giudice et al. on the CBCT assessment of radicular volume loss following TB RME highlighted that this treatment causes root volume loss of posterior teeth, with the first molars representing the teeth mostly affected by radicular resorption.

In recent years, bone-borne expansion devices have been widely used by orthodontists to reduce the undesirable effects of conventional expansion on anchorage teeth. In BB RME forces are directly applied to the palatal bone to maximize the skeletal orthopedic effect while minimizing dental side-effects. According to the systematic review by Krusi et al., bone-borne RME is associated with greater suture opening compared to tooth-borne RME, with no significant differences in term of tooth inclination, nasal cavity width and root resorption.

To date, researchers have assessed RR following orthodontic treatment using different methods, including two-dimensional radiographs, CBCT, microtomography (micro-CT), histologic examinations and scanning electron microscopy (SEM). According to Wang et al., CBCT technology offers high accuracy in assessing volumetric measurements of teeth and root resorption. Furthermore, CBCT is a less invasive method when compared to SEM and histology, which typically require the extraction of the assessed teeth.

Previous studies have investigated the linear changes in root length of maxillary permanent first molars after tooth-borne and bone-borne RME. Furthermore, other studies have conducted a CBCT three-dimensional volumetric assessment of root resorption in tooth-borne RME treatment protocols. However, when comparing the effects of tooth-borne vs bone-borne RME, only two previous studies have conducted a volumetric assessment of ERR.

The objective of this study was to compare the effects of tooth-borne (hyrax) and computer-guided miniscrew-supported rapid maxillary expansion appliances (supported by 2 or 4 miniscrews) on root volume changes of maxillary permanent first molars following the active expansion phase.

The null hypotheses were that no statistically significant changes in root volume of maxillary permanent first molars after RME would be observed within each group (intra-group evaluation) and that no statistically significant differences would be observed between the three treatment protocols (inter-group evaluation).

The present study was conducted at the Department of Orthodontics of Sapienza University of Rome involving the comparative assessment of the effects of tooth-borne and bone-borne expanders. The informed consent including details of the study's content, risks and benefits was obtained by the parents or guardians. The study was assessed and approved by the ethics committee (reference number #5951).

The sample consisted of 21 subjects (13 females, 8 males) with a mean age of 11.8 years (SD 0.79 years). The patients were randomly assigned to 3 groups according to the appliance device used for the expansion: 7 subjects were treated with the tooth-borne hyrax appliance (group TB), 7 subjects were treated with a bone-borne computer-guided expander supported by 4 miniscrews (group BB4) and 7 subjects were treated with a bone-borne computer-guided expander supported by 2 miniscrews (group BB2). The randomization of the patients in the treatment groups was performed using Clinstat statistical software (Martin Bland, York, United Kingdom).

All patients underwent CBCT examinations before the application of the RME device (T0) and post-treatment, after the 6-month retention period (T1). The exposure settings were as follows: 10 mA, 90 kV, total scanning time of 15.0 seconds, effective radiation time of 4.0 seconds, voxel size of 0.2 mm, scanning area of 14 x 16.5 cm, and an effective radiation dose of approximately 524 mGy/cm2.

The CBCT images analyzed in this study were not acquired specifically for this research but were part of an ongoing prospective randomized clinical trial aimed at evaluating the skeletal and dentoalveolar effects of three different orthodontic devices. The imaging protocol was established in accordance with ethical guidelines and was approved by the relevant institutional review board.

The T0 and T1 CBCT records of patients included in this study were digitally assessed to determine the root volume changes of maxillary permanent first molars in the three dimensions. Information regarding the structural characteristics of the RME appliances and the clinical protocol are reported as follows. In the TB group, the tooth-borne hyrax appliance was designed with bands on the maxillary first molars; in the BB4 group, the bone-borne expander was supported by 4 miniscrews inserted both in paramedian and parapalatal position of the palatal vault; in the BB2 group, the bone-borne expander was supported by 2 miniscrews inserted in the paramedian region of the palate. The same type of expansion screw and expansion protocol were used in all groups. Specifically, a 10mm hyrax click screw (Dentaurum, Bologna, Italy) was activated by 4 quarter-turns on the first day and by 3 quarter-turns per day during the active phase of treatment (0.20mm per turn, 0.6mm daily) until an 8mm screw opening was achieved.

The following method was implemented to allow the digital analysis of root volume changes of maxillary permanent first molars following the active expansion phase in the treatment groups:

1. DICOM files of pre-treatment (T0) and post-treatment (T1) CBCTs were uploaded to Mimics Medical Software (Materialise, vr. 19.0, Leuven, Belgium);
2. After uploading the DICOM files, 3D model templates of the dental and bone anatomy were created for each patient, setting a minimum threshold value of 700HU and a maximum threshold value of 3095HU with the purpose of achieving an accurate evaluation of dental root volume (Figure1);
3. STL files generated in Mimics Medical Software were exported to Autodesk Meshmixer (Autodesk Inc); the 3D models of each investigated tooth (right maxillary permanent first molar and left maxillary permanent first molar, pre-treatment and post-treatment) were isolated from the surrounding anatomical structures (Figure 2);
4. The three-dimensional images of the assessed teeth were individually saved as STL files and re-imported into the Mimics Medical Software;
5. Using the function offered by Mimics Medical Software, the volume of each investigated tooth was assessed in mm3.

Statistical Analysis Descriptive statistics (mean, standard deviation, minimum, maximum,) were used. The ratio between the mean △ volume and mean volume at T0 was calculated for each tooth in all treatment groups and expressed as a percentage. All data were recorded in an Excel database (Microsoft Corporation, 2018). Data analysis was performed using statistical software (IBM SPSS Statistics, version 25.0). To test the research hypotheses, given the small number of participants, non-parametric tests were chosen. The Wilcoxon test was used to determine whether the values recorded at T1 significantly differed from those recorded at T0 within each group. To assess whether the treatment protocol influenced the values of the dependent variable, a group comparison was conducted using the Kruskal-Wallis test. Results were considered significant for a p-value < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian children in late mixed dentition or permanent dentition,
* unilateral or bilateral transverse maxillary deficiency of at least 8 mm,
* no previous orthodontic treatment,
* good oral hygiene,
* completion of apexification of permanent first molars,
* availability of adequate pre-treatment and post-retention CBCT records

Exclusion Criteria:

* any systemic syndrome
* acute oral infections

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
root volume changes of maxillary permanent first molars following the active expansion phase. | up to 14 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial Surgery, Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No